CLINICAL TRIAL: NCT00198991
Title: German Multicenter Study for Treatment Optimisation in Acute Lymphoblastic Leukemia in Adults and Adolescents Above 15 Years (Amend 3) (GMALL 07/2003)
Brief Title: German Multicenter Trial for Treatment of Newly Diagnosed Acute Lymphoblastic Leukemia in Adults (07/2003)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Nicola Goekbuget, Principal Investigator, Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMALL01
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Adult Acute Lymphocytic Leukemia
Keywords: ALL; Treatment; de novo; Minimal residual disease; Adult
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — Cyclophosphamide; Dexamethasone; Vincristine; Daunorubicin; Asparaginase; pegaspargase; Methotrexate; Cytarabine; Mercaptopurine; Granulocyte Colony-Stimulating Factor; Vindesine; Etoposide; etoposide phosphate; Prednisolone; Doxorubicin; Thioguanine; Teniposide; Stem Cell Transplantation; Idarubicin; fludarabine; Cladribine

ARMS (1):
- All patients (Experimental): All patients are treated upfront according to one arm
  Interventions: Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Vincristine; Drug: Daunorubicin; Drug: Asparaginase; Drug: Methotrexate; Drug: Cytarabine; Drug: Mercaptopurine; Drug: G-CSF; Drug: Vindesine; Drug: Etoposide; Drug: Prednisolone; Drug: Adriamycin; Drug: Thioguanine; Drug: Teniposide; Procedure: CNS irradiation; Procedure: Mediastinal Irradiation; Procedure: Stem cell transplantation (SCT); Drug: Idarubicin; Drug: Fludarabine; Drug: Cladribine

INTERVENTIONS:
Drug: Cyclophosphamide — Cytostatic drug
Drug: Dexamethasone — Antileukemic drug
Drug: Vincristine — Cytostatic drug
Drug: Daunorubicin — Cytostatic drug
Drug: Asparaginase — Cytostatic drug
  Other Names: Pegylated Asparaginase
Drug: Methotrexate — Cytostatic drug
Drug: Cytarabine — Cytostatic drug
Drug: Mercaptopurine — Cytostatic drug
Drug: G-CSF — Growth factor
Drug: Vindesine — Cytostatic drug
Drug: Etoposide — Cytostatic drug
  Other Names: Etoposide Phosphate
Drug: Prednisolone — Antileukemic drug
Drug: Adriamycin — Cytostatic drug
Drug: Thioguanine — Cytostatic drug
Drug: Teniposide — Cytostatic drug
Procedure: CNS irradiation — Cytostatic drug
Procedure: Mediastinal Irradiation — Irradiation
Procedure: Stem cell transplantation (SCT) — Stem cell transplantation
Drug: Idarubicin — Cytostatic drug
Drug: Fludarabine — Cytostatic drug
Drug: Cladribine — Cytostatic drug

SUMMARY:
The study evaluates the efficacy and tolerability of an intensified induction and consolidation therapy. Thereafter patients receive individualised treatment stratified according to relapse risk with stem cell transplantation for patients with high and very high risk of relapse. Patients with standard risk receive further consolidation and reinduction chemotherapy. In parallel minimal residual disease (MRD) is evaluated. After six months and one year the decision on intensification or discontinuation of therapy is made based on the results of MRD evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia (pro-B, common, pre-B, early T, thymic T, mature T)
* Age 15-65 yrs (*55-65 years if biologically younger according to general condition)
* Written informed consent

Exclusion Criteria:

* Severe comorbidity or leukemia associated complications
* Late relapse of pediatric ALL or ALL as second malignancy
* Cytostatic pre-treatment
* Pregnancy
* Severe psychiatric illness or other circumstances which may compromise cooperation of the patient
* Participation in other clinical trials interfering with the study therapy

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1883 (Actual)
Dates: Start 2003-04 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2013-06-30 (Actual)

PRIMARY OUTCOMES:
Remission rate | day 46
  Rate of patients with complete remission
Remission duration | up to 10 years
  Rate and probability of patients with ongoing remission after prior achievement of remission
Disease free survival | up to 10 years
  Rate and probability of patients remaining disease free i.e without relapse, death in CR or secondary malignancy
Overall survival | up to 10 years
  Rate and probability of patients remaining alive

SECONDARY OUTCOMES:
Realisation of Stem cell transplantation (SCT) | up to 10 years
  Rate of patients receiving an SCT
Toxicity according to WHO/CTCAE | after each cycle up to 2.5 years
  Rate of adverse events according to WHO/CTCAE (cycle duration in this complex protocol is variable and cannot be specified)
Response assessment based on MRD | up to 5 years
  Rate of MRD response after specific cycles

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hoelzer, MD,PhD, Study Chair — University Hospital of Frankfurt, Medical Dept. II
Locations (1):
- University of Frankfurt, Medical Dept. II, Frankfurt, Germany

REFERENCES:
- [Derived] Kobitzsch B, Gokbuget N, Schwartz S, Reinhardt R, Bruggemann M, Viardot A, Wasch R, Starck M, Thiel E, Hoelzer D, Burmeister T. Loss-of-function but not dominant-negative intragenic IKZF1 deletions are associated with an adverse prognosis in adult BCR-ABL-negative acute lymphoblastic leukemia. Haematologica. 2017 Oct;102(10):1739-1747. doi: 10.3324/haematol.2016.161273. Epub 2017 Jul 27. PMID 28751559
- [Derived] Herold T, Schneider S, Metzeler KH, Neumann M, Hartmann L, Roberts KG, Konstandin NP, Greif PA, Braundl K, Ksienzyk B, Huk N, Schneider I, Zellmeier E, Jurinovic V, Mansmann U, Hiddemann W, Mullighan CG, Bohlander SK, Spiekermann K, Hoelzer D, Bruggemann M, Baldus CD, Dreyling M, Gokbuget N. Adults with Philadelphia chromosome-like acute lymphoblastic leukemia frequently have IGH-CRLF2 and JAK2 mutations, persistence of minimal residual disease and poor prognosis. Haematologica. 2017 Jan;102(1):130-138. doi: 10.3324/haematol.2015.136366. Epub 2016 Aug 25. PMID 27561722
- [Derived] Topp MS, Gokbuget N, Zugmaier G, Degenhard E, Goebeler ME, Klinger M, Neumann SA, Horst HA, Raff T, Viardot A, Stelljes M, Schaich M, Kohne-Volland R, Bruggemann M, Ottmann OG, Burmeister T, Baeuerle PA, Nagorsen D, Schmidt M, Einsele H, Riethmuller G, Kneba M, Hoelzer D, Kufer P, Bargou RC. Long-term follow-up of hematologic relapse-free survival in a phase 2 study of blinatumomab in patients with MRD in B-lineage ALL. Blood. 2012 Dec 20;120(26):5185-7. doi: 10.1182/blood-2012-07-441030. Epub 2012 Sep 28. PMID 23024237
- [Derived] Gokbuget N, Stanze D, Beck J, Diedrich H, Horst HA, Huttmann A, Kobbe G, Kreuzer KA, Leimer L, Reichle A, Schaich M, Schwartz S, Serve H, Starck M, Stelljes M, Stuhlmann R, Viardot A, Wendelin K, Freund M, Hoelzer D; German Multicenter Study Group for Adult Acute Lymphoblastic Leukemia. Outcome of relapsed adult lymphoblastic leukemia depends on response to salvage chemotherapy, prognostic factors, and performance of stem cell transplantation. Blood. 2012 Sep 6;120(10):2032-41. doi: 10.1182/blood-2011-12-399287. Epub 2012 Apr 4. PMID 22493293
- [Derived] Gokbuget N, Kneba M, Raff T, Trautmann H, Bartram CR, Arnold R, Fietkau R, Freund M, Ganser A, Ludwig WD, Maschmeyer G, Rieder H, Schwartz S, Serve H, Thiel E, Bruggemann M, Hoelzer D; German Multicenter Study Group for Adult Acute Lymphoblastic Leukemia. Adult patients with acute lymphoblastic leukemia and molecular failure display a poor prognosis and are candidates for stem cell transplantation and targeted therapies. Blood. 2012 Aug 30;120(9):1868-76. doi: 10.1182/blood-2011-09-377713. Epub 2012 Mar 22. PMID 22442346
- [Derived] Burmeister T, Meyer C, Schwartz S, Hofmann J, Molkentin M, Kowarz E, Schneider B, Raff T, Reinhardt R, Gokbuget N, Hoelzer D, Thiel E, Marschalek R. The MLL recombinome of adult CD10-negative B-cell precursor acute lymphoblastic leukemia: results from the GMALL study group. Blood. 2009 Apr 23;113(17):4011-5. doi: 10.1182/blood-2008-10-183483. Epub 2009 Jan 14. PMID 19144982